CLINICAL TRIAL: NCT06322992
Title: App-Assisted Day Reconstruction to Reduce Treatment Burden and Logistic Toxicity in Cancer Patients - Aim 3
Status: Completed | Type: Observational
Sponsor: Daynamica, Inc. (Industry)
Collaborators: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: R41CA271962 (NIH)
Record Dates: First submitted 2024-03-13; First posted 2024-03-21 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-05

CONDITIONS: Cancer
Keywords: Logistic Toxicity; Time Toxicity
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cancer Patients Undergoing Treatment: The investigators will recruit 60 diverse cancer patients from the statewide M Health Fairview system to participate in month-long feasibility tests. The enrolled participants will be asked to: 1) Install the prototype app from the Google Play or Apple App Store on their smartphone (the investigators will provide a smartphone with the app pre-installed to participants who do not own one); 2) Carry the smartphone for 30 consecutive days while outside the home; 3) Keep smartphone location and motion services active; 4) Confirm and correct (if needed) smartphone-detected activities and trips; 5) Use the app interface to provide additional information on treatment-related activities and trips along with well-being ratings; and 6) Review a logistic toxicity summary report that will be available within the app towards the end of the field test.

SUMMARY:
The goal of this observational study is to develop a mobile app for cancer patients undergoing treatments. In Aim 3, patients will rate the quality of the app using the Mobile App Rating Scale (MARS) and their satisfaction with the three key app features. The outcome of this project will be a final prototype app with 70% of patients indicating an overall MARS score of 4.0 or more and satisfaction with the three features.

DETAILED DESCRIPTION:
Each year, more than 1.7 million new cancer patients in the U.S. undergo intense, multimodal treatments that that create numerous logistical challenges in managing treatment and everyday life priorities. In the current cancer care system, "logistic toxicity"-the toxic effects imposed by the logistical burden of carrying out cancer treatment-related tasks on patient well-being-has been largely unmeasured and unaddressed. Current methods for measuring logistic toxicity generate retrospective assessments intended for researchers. They do not offer timely information that empower patients to solicit assistance from care providers, employers, family, and friends. Nor do they empower providers to explore the increasingly available treatment options for patient- centered cancer care. This proposal aims to apply a new method-app-assisted day reconstruction-to develop the first digital health tool to enable remote patient monitoring of logistic toxicity, which is the necessary first step towards developing effective care interventions for addressing it.

Our product is both conceptually and technically innovative. Conceptually, the investigators apply the day reconstruction method-a method initially created by well-being researchers for collecting more accurate data on daily life experiences-to collect activity engagement and well-being information related to cancer treatment tasks. Technically, the investigators leverage the existing patented technology and new machine learning techniques to enable novel integration of objective mobile sensing with subjective patient input. Mobile sensing and machine learning will constitute the "assist" that the app provides for day reconstruction in relation to logistic toxicity, significantly reducing recall errors and the need for manual input. The "assist" will also prompt patients to provide information such as subjective well-being ratings that are not detectable by mobile sensing or machine learning, generating more accurate and comprehensive measures of logistic toxicity than existing methods.

The project has three specific aims, including (1) an initial system design based upon input from cancer patients and cancer care stakeholders, (2) prototype development and initial tests, and (3) field tests of the app among 60 diverse patients undergoing treatment for cancer. In Aim 3, patients will rate the quality of the app using the Mobile App Rating Scale (MARS) and their satisfaction with the three key app features: 1) the app's ability to capture out-of-home treatment-related activities and trips, 2) the ease of the interface for inputting home-based treatment-related activities and well-being ratings, and 3) the usefulness of the logistic toxicity summary report. The outcome of this project will be a final prototype app with 70% of patients indicating an overall MARS score of 4.0 or more and satisfaction with the three features. In Phase II, the team will test the efficacy of the app-both separately and in conjunction with care coordination, telemedicine, and home-based treatments-in reducing logistic toxicity and improving treatment outcomes in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients undergoing treatments

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 60 diverse cancer patients, oversampling socio- economically disadvantaged populations
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
APP satisfaction | March 2024 - May 2025
  The investigators will recruit 60 diverse cancer patients, oversampling socio- economically disadvantaged populations, to conduct month-long usability tests followed by exit surveys. Patients will rate satisfaction with the three app features developed in Aim 2 using the 5-point Likert scale. The Aim 3 milestone will be 70% of patients indicating satisfied/very satisfied with each of the three features.
APP rating | March 2024 - May 2025
  The investigators will recruit 60 diverse cancer patients, oversampling socio- economically disadvantaged populations, to conduct month-long usability tests followed by exit surveys. Patients will rate the overall app quality using the Mobile App Rating Scale (MARS) that encompasses engagement, functionality, aesthetics, information, and subjective quality. The Aim 3 milestone will be an overall MARS score of 4.0 or above.

CONTACTS AND LOCATIONS:
Overall Officials: Yingling Fan, Principal Investigator — Daynamica, Inc.
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No